CLINICAL TRIAL: NCT03505125
Title: A Non-Interventional Observational Study of Pegvaliase-Naïve Adults With Phenylketonuria (PKU): Concept Elicitation and Cognitive Interviews
Brief Title: A Non-Interventional Interview Study of Phenylketonuria (PKU) Adults
Acronym: 165-901
Status: Completed | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 165-901
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Phenylketonuria (PKU)
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PKU Patients: Adults with PKU will be interviewed about the symptoms and impacts of PKU.
- Observers: Close friends and family members of adults with PKU will be interviewed about the behaviors they have observed in adults with PKU
- Clinical Experts: Experienced, practicing clinicians currently treating adults with PKU will be interviewed about the symptoms and impacts of PKU on their patients.

SUMMARY:
The 165-901 study is designed to identify the appropriate tools for use in future interventional studies on the neurocognitive effects of pegvaliase on adults with PKU.

DETAILED DESCRIPTION:
Clinical studies have suggested that treatment with pegvaliase results in lowering of blood Phenylalanine levels in adults with Phenylketonuria (PKU). Because these individuals often exhibit inattention and mood difficulties, and blood Phe concentration affects cognition and mood, life-long blood Phe control with pegvaliase may improve cognitive abilities and emotional and mental health in patients with PKU. In order to adequately quantify potential pegvaliase treatment impact on cognition and mood, it is necessary to employ clinical outcome assessments (COAs) that are fit for purpose and that comprehensively address concepts important, relevant, and meaningful to PKU patients. This is an observational study to identify symptom, function, and health-related quality of life (HRQoL) concepts of interest (COIs) to patients with PKU and to seek additional patient, observer, and expert input on the appropriateness of concepts of BioMarin's proposed COAs for use in future efficacy trials in PKU.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible to participate in this study must meet all of the following criteria:

1. ≥18 and ≤70 years of age at the time of consent;
2. Clinically-confirmed diagnosis of Phenylketonuria (PKU);
3. Blood Phe test completed within eight weeks prior to screening date or blood Phe test completed within eight weeks post screening date;
4. Able to read, understand, and speak fluently the language(s) of their designated country sufficiently to participate in an interview and/or complete all assessments;
5. Willing and able to participate in a telephone interview lasting approximately 90 minutes;
6. Willing to be audio-recorded during the interview session;
7. Willing and able to provide written informed consent indicating that they understand the purpose and procedures required for the study and are willing to participate.

Exclusion Criteria:

Patients meeting any of the following criteria will not be included in the study:

1. Currently pregnant;
2. Current or previous exposure to pegvaliase treatment or participation in a pegvaliase clinical trial;
3. Has a significant cognitive impairment, hearing difficulty, visual impairment, acute psychopathology, medical condition, or insufficient knowledge of the interview language that, in the opinion of the investigator or interviewer, would interfere with his or her ability to provide written consent and participate/complete an interview.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Individuals with PKU ≥18 years to ≤ 70 years of age who are naïve to pegvaliase
  2. Observers ≥18 years of an individual with PKU ≥18 years to ≤ 70 years of age who are naïve to pegvaliase
  3. Clinical experts currently treating PKU adults
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2018-03-31 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
PKU Symptom Survey | 15 minutes
  60 item survey asking patients, observers and clinical experts about the symptoms and behaviors associated with PKU and changes in Phe level.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (14):
- United States (4):
  - University of Florida, Gainesville, Florida
  - Emory University Department of Human Genetics, Decatur, Georgia
  - Ann and Robert H Lurie Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
- Adult Metabolic Diseases Clinic, Vancouver General Hospital, Vancouver, British Columbia, Canada
- France (2):
  - Necker Children's Hospital, Paris, Cedex 15
  - Bretonneau Hospital, Internal Medicine Department, Tours, Cedex 9
- Germany (2):
  - University Klinik Jena, Klinik für Neuropädiatrie, Jena, Thuringia
  - Rheumatology Unit, Clinic for Inborn Errors of Metabolism, Leipzig
- Italy (2):
  - Hospital of Padova, Padua
  - Umberto I Polyclinic of Rome, Roma
- Turkey (Türkiye) (2):
  - Hacettepe University, Ankara
  - Ege University School of Medicine, Izmir
- National Hospital for Neurology and Neurosurgery, London, England, United Kingdom